CLINICAL TRIAL: NCT00436137
Title: Improving Followup of Positive Fecal Occult Blood Tests
Brief Title: Improving Followup of Abnormal Colon Cancer Screening Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Vanguard Medical Associates (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Thomas Sequist, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Sequist Colorectal Cancer
Record Dates: First submitted 2007-02-14; First posted 2007-02-16 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Fecal occult blood test; Abnormal test result; Missed diagnosis; Delayed diagnosis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients will receive a mailing recommending colonoscopy, followed by a telephone outreach
  Interventions: Behavioral: Patient mailing

INTERVENTIONS:
Behavioral: Patient mailing — Patient will receive a mailing recommending colonoscopy, followed by telephone outreach

SUMMARY:
The purpose of this study is to determine whether direct mailings to patients with positive fecal occult blood tests can increase rates of performing followup colonoscopy.

DETAILED DESCRIPTION:
Screening programs using the fecal occult blood test (FOBT) have demonstrated a significant reduction in colorectal cancer mortality, although only when accompanied by a complete diagnostic evaluation of the colon in the setting of a positive result. 90% of patients with a positive FOBT result have completed a subsequent colonoscopy within Harvard Vanguard Medical Associates. This project will use a pre-post study design to increase the rate of followup colonoscopy in the setting of positive FOBT results. Patients in the intervention group will receive a personalized mailing highlighting their positive result and need for colonoscopy, followed by telephone outreach from a centralized gastroenterology scheduling office. The primary outcome will be the performance of colonoscopy, however we will also perform chart reviews to identify predictors of completing appropriate followup.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive fecal occult blood test during 2004, 2005, and 2006; and no colonoscopy following this test result

Exclusion Criteria:

* Patients with active cardiopulmonary disease or limited life expectancy due to severe illness such as malignancy
* Colonoscopy within 5 years prior to positive fecal occult blood test
* Age > 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Performance of colonoscopy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Sequist, MD, MPH, Principal Investigator — Harvard Vanguard Medical Associates
Locations (1):
- Harvard Vanguard Medical Associates, Newton, Massachusetts, United States